CLINICAL TRIAL: NCT05091138
Title: Are Adductor Canal Blocks With Bupivacaine and Added Magnesium Better at Managing Post-operative Pain Than Adductor Canal Blocks With Bupivacaine and Added Buprenorphine in Patients Undergoing Same-day Discharge Total Knee Arthroplasty?
Brief Title: Are Adductor Canal Blocks With Bupivacaine and Added Magnesium Better at Managing Post-operative Pain Than Bupivacaine and Added Buprenorphine in Patients Undergoing Same-day Discharge Total Knee Arthroplasty?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Sandeep Krishnan, Associate Professor of Anesthesiology, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Mg versus Buprenorphine in TKA
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Post-operative Pain, Acute; Opioid Use
Keywords: Same-day discharge total knee arthroplasty; Magnesium; Adductor canal block; Post-operative opioid consumption; Post-operative pain management
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mg and Bupivacaine (Active Comparator): Patients in this arm (selected randomly) will receive an ultrasound-guided adductor canal block (ACB) with 30cc of 0.25% bupivacaine and 150mg of Mg.
  Interventions: Drug: Adding Magnesium as an adjuvant to Bupivacaine in the adductor canal block (ACB) for same-day discharge total knee arthroplasty
- Buprenorphine and Bupivacaine (Active Comparator): Patients in this arm (selected randomly) will receive an ultrasound-guided adductor canal block (ACB) with 30cc of 0.25% bupivacaine and 300 mcg of buprenorphine.
  Interventions: Drug: Adding Buprenorphine as an adjuvant to Bupivacaine in the adductor canal block (ACB) for same-day discharge total knee arthroplasty

INTERVENTIONS:
Drug: Adding Magnesium as an adjuvant to Bupivacaine in the adductor canal block (ACB) for same-day discharge total knee arthroplasty — Post-operatively all patients will have an ultrasound-guided adductor canal block (ACB) with 30cc of 0.25% bupivacaine. Half of the patients (selected randomly using random number table) will receive 150mg of magnesium sulfate in the block and the other half will receive 300 mcg of buprenorphine in the block.
  Arms: Mg and Bupivacaine
Drug: Adding Buprenorphine as an adjuvant to Bupivacaine in the adductor canal block (ACB) for same-day discharge total knee arthroplasty — Post-operatively all patients will have an ultrasound-guided adductor canal block (ACB) with 30cc of 0.25% bupivacaine. Half of the patients (selected randomly using random number table) will receive 150mg of magnesium sulfate in the block and the other half will receive 300 mcg of buprenorphine in the block.
  Arms: Buprenorphine and Bupivacaine

SUMMARY:
The purpose of this study is to compare the use of magnesium and bupivacaine to buprenorphine and bupivacaine in post-operative adductor canal blocks (ACB); the study will determine if one combination can result in decreased opioid consumption and improved pain management for patients after same-day discharge total knee arthroplasty (TKA) .

The investigators will assess whether the addition of magnesium to bupivacaine will decrease visual analog scale (VAS) pain scores, decrease post-operative total opioid consumption (oral morphine equivalents), decrease the incidence of post-operative nausea and vomiting (PONV), and improve patient satisfaction in comparison to when buprenorphine is added to bupivacaine.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is one of the most common elective surgical procedures in the United States . The number of TKA procedures has doubled in each of the past two decades and is expected to top 3.4 million per year in the United States by 2030.

Within the last 10-15 years significant changes have taken place in the anesthetic management of patients undergoing total knee arthroplasty (TKA). In the past, the majority of patients underwent general anesthesia and were managed post-operatively with a PCA (patient controlled analgesia) pump.

More recently anesthesiologists have begun to use neuraxial anesthesia (spinal anesthesia) combined with regional anesthesia (peripheral nerve block (PNB)) techniques combined with monitored anesthesia care (MAC) for many of these surgeries.

Regional anesthesia is used to block the sensation in a specific part of body during and after surgery. It offers numerous advantages over conventional general anesthesia, including faster recovery time, fewer side effects, no need for an airway device during surgery, and a dramatic reduction in post-surgical pain and reduction in opioid use following surgery. The use of local anesthetic peripheral nerve blocks for surgical anesthesia and postoperative pain management has increased significantly with the advent of ultrasound-guided techniques.

However, the duration of traditional amide-based and ester-based regional anesthesia is normally limited to only a few hours. Techniques including continuous catheter placement or serial injections can be used to enhance the duration and effect of regional anesthesia for postoperative pain control. But these approaches can increase the risk of infection, toxicity, and cost. Therefore, alternative methods of extending the clinical duration of nerve blocks have been a topic of significant interest.

The purpose of this study is to determine whether the addition of magnesium to bupivacaine for the post-operative adductor canal blocks can decrease opioid consumption and improve pain management for patients after total knee arthroplasty (TKA) versus adding buprenorphine to bupivacaine for the blocks.

The investigators will assess whether the addition of magnesium will decrease visual analog scale (VAS) pain scores, decrease post-operative total opioid consumption (oral morphine equivalents), decrease the incidence of post-operative nausea and vomiting (PONV), and improve patient satisfaction in comparison to when buprenorphine is administered instead.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral primary total knee arthroplasty with spinal anesthetic and MAC followed by a unilateral adductor canal block with ultrasound guidance.

Exclusion Criteria:

* Patients on chronic anticoagulation upon admission
* Patients with significant genetic or acquired clotting/bleeding disorders (hemophilia, DIC, etc.) or significant platelet dysfunction
* Patients with prior back surgery or leg surgery that precludes spinal or regional anesthesia
* Infection at sites for regional/spinal anesthesia
* Allergy to local anesthetics

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Total opioid consumption (oral morphine equivalents) in the first 24 hours after surgery | The first 24 hours after surgery
  Measuring the post surgical total opioid consumption in the first 24 hours after surgery by calculating oral morphine equivalents (mg)
Total opioid consumption (oral morphine equivalents) in the second 24 hours after surgery | The second 24 hours after surgery
  Measuring the post surgical total opioid consumption in the second 24 hours after surgery by calculating oral morphine equivalents (mg)
Visual analog scale (VAS) pain score at 24 hours after surgery | 24 hours after surgery
  Determining pain scores using Visual analog scale (VAS) at 24 hours after surgery (0-10, Higher scores mean worse outcome)
Visual analog scale (VAS) pain score at 48 hours after surgery | 48 hours after surgery
  Determining pain scores using Visual analog scale (VAS) at 48 hours after surgery (0-10, Higher scores mean worse outcome)

SECONDARY OUTCOMES:
Percentage of incidence of post-operative nausea/ vomiting in first 48 hours after surgery | First 48 hours after surgery
  The incidence of nausea or vomiting in the first 48 hours after surgery is recorded
Overall patient satisfaction in first 48 hours after surgery | First 48 hours after surgery
  Patient satisfaction scores averaged over the first 48 hours after surgery (0-10, higher scores are better)

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph Mercy Oakland Hospital, Pontiac, Michigan, United States

IPD SHARING:
Plan to Share IPD: No